CLINICAL TRIAL: NCT03859154
Title: Waveform Analysis In Snakebite Victims With Hematotoxicity
Acronym: WISH
Status: Completed | Type: Observational
Sponsor: Jubilee Mission Medical College and Research Institute (Other)
Responsible Party: Principal Investigator, Siju V Abraham, MD, Assistant Professor in the Department of Emergency Medicine, Jubilee Mission Medical College and Research Institute
Other Study IDs: 05/19/IEC/JMMC&RI; U1111-1229-0385 (Other: World Health Organisation)
Record Dates: First submitted 2019-02-26; First posted 2019-03-01 (Actual); Last update posted 2023-07-17 (Actual); Status verified 2023-07

CONDITIONS: Snakebite; Coagulopathy, Consumption
MeSH Terms: conditions — Snake Bites; Disseminated Intravascular Coagulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Viper bite victims: Snakebite victims in whom the snake has been brought and positively identified as Viperidae AND simultaneous aPTT has been sent AND consenting to be part of the study
- Nonvenomous snakebite: age and gender matched victims of snake bite in whom the culprit snake brought along has been identified as a non venomous one.
  AND consenting to be part of the study

SUMMARY:
In hematotoxic snakebites, due to the lack of a better alternative, 20 minute whole blood clotting test (20'WBCT) or Clotting time remains the standard test in developing countries even though its reliability and sensitivity has been shown to be low.

Activated partial thromboplastin time (aPTT) based Clot Waveform Analysis (CWA) is an optic absorbance assay that can be used as a global clotting test.

It essentially detects the change in colour of the plasma as coagulation progresses and quantifies the change in the form of a waveform.

In this study, the investigators intend to study prospectively the behaviour of clot wave (CW) in hematotoxic bites.

A pilot observational study was initially conducted (IEC Ref No. 42/16/IEC/JMMC and RI) and CWA showed changes which provided information earlier than the conventional coagulation studies in the snakebite victims studied.

While aPTT or WBCT reflects clotting time, CWA conveys the dynamic process of clot formation. CWA may reveal disorders of clotting in snakebite victims before the conventional tests become abnormal.

Here the investigators aim to study the changes in CWA in snakebite victims who develop coagulation disorders in blood

DETAILED DESCRIPTION:
Viperidae bites are quite common in India and are notorious to cause hematotoxicity.

In hematotoxic bites, the test recommended to ascertain the development of coagulopathy is a whole blood clotting test (WBCT) as per the current guidelines.

Eventhough the reliability and sensitivity of WBCT has been shown to be low, it still remains the standard test.

There exists a need to explore other coagulation studies in snakebite to look for a better and efficient alternative.

Clot waveform analysis (CWA) is an activated partial thromboplastin time (aPTT)-based optic absorbance assay that can be used as a global clotting test.

It has been shown useful in identifying disseminated intravascular coagulation (DIC) in sepsis with high specificity (97.6%) and sensitivity (98%), and the test is recommended by the British Committee for Standards in Hematology guidelines for the diagnosis and treatment of DIC.

CWA is based on the traditional aPTT assay. On assessing aPTT with light transmission, a change in the light absorbance is observed as the clot stabilizes by fibrin polymerization.

Plotting the milliabsorbance (mAbs) of the sample to time, a curve is obtained which reflects the optical profile that is generated as a clot is formed.

This tracing against time gives a qualitative assessment of fibrin polymerization.

The delta in absorbance (dAbs) is based on the change in mAbs value from the baseline to the endpoint (plateau) along the Y-axis of the clot curve. The dAbs values of <100 mAbs denote low fibrinogen samples

The normal clot waveform has five main phases: delay, baseline, acceleration, deceleration, and end point.

The "delay" period begins at 0 and precedes the "baseline." which denotes the mixing of the reagents and system optimization of light intensity.

The "baseline" is the portion of the curve which appears after all reagents have been added to the time and the clot formation begins.

The aPTT value is noted at this point (vertical red line). The "acceleration" phase denotes fibrin clot formation, whereas "deceleration" denotes decreasing rate of clot formation.

There are two more curves that are plotted in CWA, the first derivative and the second derivatives. They are both derivatives of the absorbance curves. The first derivative reflects the coagulation velocity, whereas the second derivative reflects the acceleration of coagulation.

The investigators in this study aim to assess the changes in the CW form in viper-envenomated victims and to compare CWA with standard tests such as prothrombin time (PT) with the international normalized ratio (INR), aPTT, clotting time (CT) (modified Lee and White method) and 20'WBCT( twenty minute whole blood clotting test)

ELIGIBILITY:
Inclusion Criteria:

-snakebite victims were activated Partial Thromboplastin Time (aPTT) sample has been sent

Exclusion Criteria:

* Not consenting to be part of the study
* OR known case of coagulation disorders
* OR chronic liver disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All victims of snakebite consenting to be part of the study presenting to the emergency department at Jubilee Mission Medical College and Research Institute Thrissur, Kerala, India
  Snake bite registry would be established All consecutive cases would be enrolled in the study if they consent to be part of it.
  Sub group analysis excluding the dry bites,would be done Sub group analysis of the victims of hematotoxic snakebite would be done
Sampling Method: Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Clot wave form 1st derivative changes | For all aPTT samples done at admission, just prior to antivenom administration, 6 hours after antivenom administration completion and 6 hours after blood product administration, upto 7 days post admission.
  Changes in the 1 st derivative
Clot wave form 2nd derivative changes | For all aPTT samples done at admission, just prior to antivenom administration, 6 hours after antivenom administration completion and 6 hours after blood product administration, up to 7 days post admission.
  Changes in the 2nd derivative
changes in delay phase, baseline, acceleration, deceleration and end point phases of CWA | For all aPTT samples done at admission, just prior to antivenom administration, 6 hours after antivenom administration completion and 6 hours after blood product administration, up to 7 days post admission.
  Changes in the predefined Clot wave segments

SECONDARY OUTCOMES:
Clotting time (CT) | For all CT samples done at admission, just prior to antivenom administration, 6 hours after antivenom administration completion and 6 hours after blood product administration, up to 7 days post admission..
  The absolute clotting time by modified lee white method done for all samples as per institutional protocol
maximum coagulation velocity | For all aPTT samples done at admission, just prior to antivenom administration, 6 hours after antivenom administration completion and 6 hours after blood product administration, up to 7 days post admission.
  maximum coagulation velocity

OTHER OUTCOMES:
sensitivity and specificity of CWA in detecting envenomation compared to 20'WBCT and MLW (Modified Lee and White) method | from admission till time of objective detection of coagulopathy, or up to 48 hours of admission, whichever is earliest
  To test how sensitive and specific changes in CWA is in detecting coagulopathy in snakebite victims compared to the World Health Organisation Recommended twenty minute whole blood clotting test and the modified lee white clotting time done as per institute protocol
correlation of CWA with serum fibrinogen levels | For all serum Fibrinogen and aPTT sample sent simultaneously upto 48 hours of admission.
  For all serum Fibrinogen and aPTT sample sent simultaneously correlation of CWA parameters with serum fibrinogen levels

CONTACTS AND LOCATIONS:
Overall Officials: Siju V Abraham, M.D, Principal Investigator — Jubilee Mission Medical College and Research Institute
Locations (1):
- Jubilee Mission Medical College and Research Institute, Thrissur, Kerala, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Abraham SV, Rafi AM, Krishnan SV, Palatty BU, Innah SJ, Johny J, Varghese S. Utility of Clot Waveform Analysis in Russell's Viper Bite Victims with Hematotoxicity. J Emerg Trauma Shock. 2018 Jul-Sep;11(3):211-216. doi: 10.4103/JETS.JETS_43_17. PMID 30429630